CLINICAL TRIAL: NCT02313376
Title: Trial to Assess the Safety, Attenuation and Immunogenicity of Genetically-attenuated p52-/p36-/sap1- Plasmodium Falciparum Parasites (GAP3KO) Administered Via Infected Anopheles Stephensi Mosquitoes to Malaria-Naïve Adults
Brief Title: Safety, Attenuation and Immunogenicity of GAP3KO Administered Via A Stephensi Mosquitoes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MC-004
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GAP3KO (Experimental)
  Interventions: Biological: GAP3KO

INTERVENTIONS:
Biological: GAP3KO — GAP3KO administered via the bite of 150-200 GAP3KO-infected A. stephensi mosquitoes under controlled conditions.

SUMMARY:
Study designed to evaluate safety and tolerability of a genetically attenuated P. falciparum (GAP3KO) that arrests early in the liver stage of the parasite life cycle. Study will also confirm the attenuation of the GAP3KO parasites using peripheral blood smears. Secondary objectives are to evaluate the humoral immune responses to GAP3KO.

DETAILED DESCRIPTION:
This single arm, open-label, phase 1 safety study is designed to evaluate the safety and tolerability of a genetically attenuated P. falciparum (GAP3KO) that arrests early in the liver stage of the parasite life cycle. The study will also confirm the attenuation of the GAP3KO parasites using peripheral blood smears. The secondary objectives of the study are to evaluate the humoral immune responses to GAP3KO.

A total of 10 healthy, malaria-naïve adult subjects will be enrolled to receive GAP3KO via the bite of 150-200 GAP3K0-infected A. stephensi mosquitoes under controlled conditions. Subjects will be evaluated for safety, reactogenicity, and signs and symptoms of malaria to confirm attenuation for 28 days, including monitoring in a hotel setting 8-18 days post GAP 3KO administration.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* No hematologic, hepatic, or renal disease
* Weight greater than 50 kg
* Assessment of Understanding completed and passed prior to enrollment
* Availability and reliable access to trial center
* Females must use two forms of pregnancy prevention

Exclusion Criteria:

* Recent (within 6 months) or planned travel to malaria endemic area
* History of confirmed malaria diagnosis
* Anticipated use of the following:

  * Investigational malaria vaccine at any time
  * Malaria chemoprophylaxis within 6 months
  * Chronic systemic immunosuppressive medications within 6 months
  * Blood products or immunoglobulin within 120 days
  * Systemic antibiotics with antimalarial effects within 30 days
  * Investigational product or vaccine within 30 days
  * Live vaccine within 28 days; killed vaccine within 14 days of GAP3KO
  * Medications known to significantly interact with chloroquine or Malarone
* History of:

  * Sickle cell trait or other hemoglobinopathies
  * Splenectomy or functional asplenia
  * Systemic anaphylaxis
  * Severe allergic reaction to mosquito bites or malaria treatment drugs
  * History of chronic or active neurologic disease
  * Cardiac disease or stroke
* Clinically significant medical condition, abnormal lab results
* Clinically significant abnormal ECG
* Moderate or high risk for coronary heart disease
* Acute illness
* Pregnant or nursing female
* HIV, Hepatitis B, or Hepatitis C
* Psychiatric condition that precludes compliance with the protocol
* Suspected or known alcohol or drug abuse
* Staff with direct involvement in conduct of the study or GAP activities

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Safety assessed by frequency of AEs, SAEs, and patent parasitemia via peripheral blood smear | 28 Days

SECONDARY OUTCOMES:
CSP antibody titer | 28 days
Percent inhibition of in vitro sporozoite | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Biomedical Research Institute Malaria Clinical Trial Center, Seattle, Washington, United States